CLINICAL TRIAL: NCT02600442
Title: Assessment of Breast Cancer Response to Neoadjuvant Anthracycline-based Chemotherapy by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) and Molecular Markers
Brief Title: Assessment of Breast Cancer Response to Neoadjuvant Anthracycline-based Chemotherapy by FDG-PET and Molecular Markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/27NICB
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Neoadjuvant Therapy; Chemotherapy; Positron-Emission Tomography; PET-CT; FDG; Fluorodeoxyglucose; Diagnosis; Prognosis; Pathological complete response; molecular biology; proliferation genes
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — somatic molecular analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- main and unique cohort
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study

SUMMARY:
A correlation between early changes in the tumor maximum standardized uptake value (SUVmax) on FDG-PET after one or two cycles of neoadjuvant chemotherapy (NAC) and the pathological response after 6 to 8 cycles has been demonstrated in several independent small series of patients.

Breast tumor proliferation status has previously been demonstrated to be a good predictive factor of response to chemotherapy. The best method for assessing proliferation status is unclear. Proportion of cells staining for nuclear Ki67 antigen is the most widely used assay for comparing the proliferation status between tumors. However major variations in analytical procedure and interpretation limited its clinical value. Taking into account the prognosis and predictive value of proliferation gene as a common "signature" in breast cancer transcriptome analysis, quantitative assessment of mRNA expression of genes involved in proliferation has been developed by the investigators team and others. The evaluation of these parameters is quantitative and reliable and can be standardized for a clinical use.

The main objective of the investigators study is to early predict pathological response to anthracycline-based neoadjuvant chemotherapy (NAC) using a combination of parameters based on FDG-PET imaging performed at baseline and after 2 cycles, and molecular markers of proliferation measured on pre-treatment biopsy (Ki67 protein level by immunohistochemistry and Ki67 mRNA level and the mRNA (messenger RNA) expression of the most pertinent genes of the Genomic Grade Index (GGI) component by RT (reverse transcriptase) - qPCR).

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Newly diagnosed invasive breast cancer
* Stage-II or stage-III
* Neoadjuvant anthracycline-based chemotherapy
* Primary breast biopsy must be available
* Non metastatic, M0
* No prior systemic therapy for the presFrance: Direction Generale de la Sante ent tumor
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures

Exclusion Criteria:

* Metastatic breast cancer
* Uncontrolled diabetes
* Limited breast cancer immediately accessible to conservative surgery and not candidate for neoadjuvant chemotherapy
* Previous homolateral breast cancer and/or contralateral breast cancer except if treated by surgery +/- radiation therapy alone without any systemic treatment
* Any surgery (not including minor procedures such as lymph node biopsy, primary tumor core biopsy, fine needle aspiration) within 12 weeks of start of study treatment; or not fully recovered from any side effects of previous procedures.
* Diagnosis of any previous malignancy within the last 5 years, except for adequately treated basal cell carcinoma, or squamous cell skin carcinoma, or in situ cervical carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage II-III Breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response to anthracycline-based neoadjuvant chemotherapy | Within the first 30 days after surgery
  * To analyze separately clinical, pathological and molecular biomarkers currently used to identify molecular breast cancer subgroups of the primary tumor that, coupled with the metabolic response, could improve early pathological prediction.
  * To analyze separately the biological, molecular, and genetic biomarkers from the study that, coupled with the metabolic response, could improve early pathological prediction.
  * To analyze separately high throughput analysis of molecular biomarkers of the primary tumor that, coupled with the metabolic response, could improve early pathological prediction.

SECONDARY OUTCOMES:
Overall Survival | 5 years
Overall Survival | 3 years
Event Free survival | 5 years
  To determine the 5 years Event free survival (EFS) rates in breast cancer patients according to PET response, biological markers and biomarkers identified with molecular high throughput analysis.
Event Free survival | 3 years
  To determine the 3 years Event free survival (EFS) rates in breast cancer patients according to PET response, biological markers and biomarkers identified with molecular high throughput analysis.
Breast Cancer specific survival | 5 years
  To determine the 5 years Breast Cancer Specific survival rates in breast cancer patients according to PET response, biological markers and biomarkers identified with molecular high throughput analysis.
Breast Cancer specific survival | 3 years
  To determine the 3 years Breast Cancer Specific survival rates in breast cancer patients according to PET response, biological markers and biomarkers identified with molecular high throughput analysis.
Pathological partial response to anthracycline-based neoadjuvant chemotherapy | Within the first 30 days after surgery
  * To analyze separately clinical, pathological and molecular biomarkers currently used to identify molecular breast cancer subgroups of the primary tumor that, coupled with the metabolic response, could improve early pathological prediction.
  * To analyze separately the biological, molecular, and genetic biomarkers from the study that, coupled with the metabolic response, could improve early pathological prediction.
  * To analyze separately high throughput analysis of molecular biomarkers of the primary tumor that, coupled with the metabolic response, could improve early pathological prediction.
Delta SUV | Within the first 20 days after the second cycle of chemotherapy
  To evaluate the correlation between baseline molecular status of proliferation and FDG uptake measured at baseline, after 2 cycles of NAC and the change (delta SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Veron, Study Chair — DRCD; Patricia de Cremoux, MD-PhD, Principal Investigator — APHP, IUH, University Paris Diderot, Paris 7, SPC; David Groheux, MD-PhD, Principal Investigator — APHP, IUH, University Paris Diderot, Paris 7, SPC
Locations (1):
- Hopital siant-Louis, Paris, Paris, France